CLINICAL TRIAL: NCT00001329
Title: Plasma Catecholamine Kinetics
Brief Title: Study of Norepinephrine Levels and Sympathetic Nervous System Activity
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 920259; 92-N-0259
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-09

CONDITIONS: Autonomic Nervous System Disease; Healthy; Hypertension
Keywords: Yohimbine; Catecholamines; Sympathoadrenal Response; Sympathetic Nervous System; Stress; Hypertension; Autonomic Failure
MeSH Terms: conditions — Hypertension; Pure Autonomic Failure

SUMMARY:
Brain and nerve cells communicate with each other by releasing and picking up chemicals called neurotransmitters. Norepinephrine is a neurotransmitter used by part of the nervous system activated during stress called the sympathetic nervous system. The sympathetic nervous system is involved with regulating blood pressure and pulse rate. Researchers believe the level norepinephrine in the blood can be used to measure activity of the sympathetic nervous system.

This study is designed to answer important questions about rates of release of norepinephrine into the blood stream, removal of released norepinephrine, and the sympathetic nervous system response to stress.

Researchers will attempt to measure levels of norepinephrine and activity of the sympathetic nervous system in patients with high blood pressure, normal patients with family histories of high blood pressure, patients taking drugs that can effect levels of norepinephrine, and patients with diseases or conditions directly affecting the sympathetic nervous system.

DETAILED DESCRIPTION:
In order to examine sympathetic nervous system function in neurocardiological disorders and catecholaminergic effects of dietary manipulations or neuropsychiatric drugs, the protocol calls for evaluations of the kinetics of 3H-norepinephrine or 3H-epinephrine in patients with hypertension, dysautonomias, or disorders thought to involve abnormal catecholaminergic function, and in normotensive normal volunteers. Apparent spillover and clearance rates are estimated based on the norepinephrine or epinephrine concentration during the infusion and their steady-state specific activities, under resting conditions and in response to physiological or pharmacological manipulations thought to affect sympathetic outflows.

ELIGIBILITY:
Must be greater than or equal to 18 years of age.

Must not be pregnant or lactating.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 1992-09; Study Completion 2002-09

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Goldstein DS, Horwitz D, Keiser HR, Polinsky RJ, Kopin IJ. Plasma l-[3H]norepinephrine, d-[14C]norepinephrine, and d,l-[3H]isoproterenol kinetics in essential hypertension. J Clin Invest. 1983 Nov;72(5):1748-58. doi: 10.1172/JCI111134. PMID 6630523
- [Background] Rea RF, Eckberg DL, Fritsch JM, Goldstein DS. Relation of plasma norepinephrine and sympathetic traffic during hypotension in humans. Am J Physiol. 1990 Apr;258(4 Pt 2):R982-6. doi: 10.1152/ajpregu.1990.258.4.R982. PMID 2331039
- [Background] Goldstein DS, Eisenhofer G, Stull R, Folio CJ, Keiser HR, Kopin IJ. Plasma dihydroxyphenylglycol and the intraneuronal disposition of norepinephrine in humans. J Clin Invest. 1988 Jan;81(1):213-20. doi: 10.1172/JCI113298. PMID 3335637